CLINICAL TRIAL: NCT00865956
Title: A Comprehensive Disease Management Program for Medically-Complex Substance Users
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Johns Hopkins University (Other)
Collaborators: Johns Hopkins Community Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00015261
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Substance-related Disorder
Keywords: disease management; substance use disorders; behavioral incentives
MeSH Terms: conditions — Substance-Related Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care Management (Experimental): Care Management plus voucher incentives for adherence to primary care appointments.
  Interventions: Behavioral: Contingency Management; Other: Case management
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Contingency Management — Rite Aid vouchers (stepped value) for reinforcement of adherence to primary care
  Arms: Care Management
Other: Case management — Nurse case manager assigned to participant
  Arms: Care Management

SUMMARY:
Disease management (DM) programs are being increasingly utilized by health plans to coordinate care, improve quality of care, and control costs in chronically ill individuals. DM programs for specific medical conditions, such as diabetes mellitus, congestive heart failure, and asthma, have demonstrated improvements in health outcomes and a number of studies have found economic benefits to these programs as well. There are fewer data evaluating multi-disease DM programs, and results have been mixed. Additionally, data on such programs specifically targeting substance-using populations are limited, although they are promising. Prior utilization and hospitalization data from Johns Hopkins Hospital, Johns Hopkins Health Care, and Priority Partners Managed Care Organization (PPMCO) suggest that a substantial portion of high-utilizing, high-cost, medically complex patients have a substance use diagnosis.

The investigators hypothesize that a comprehensive DM program for medically-complex substance users with a history of hospitalization, consisting of intensive nurse case management along with behavioral incentives to reinforce engagement in primary care, can decrease inpatient days and costs, as well as improve outcomes for substance use, depression, and physical and mental functioning. The investigators will compare the case management/behavioral incentives intervention to usual care among a group of medically-complex, substance-using, PPMCO enrollees. Usual care will include access to all existing Priority Partners care management programs, and usual The investigators believe that this research will make an important contribution to the development of models of chronic care that improve health and promote the best use of health care resources. Additionally, the investigators believe this project will promote the study and development of systems to improve the health of substance-using adults, an underserved and often marginalized group.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Continuous enrollment in Priority Partners MCO for past 12 months
* Primary care site East Baltimore Medical Center (EBMC)
* PPMCO substance abuse flag other than nicotine only within past 24 months

Exclusion Criteria:

* currently enrolled in PPMCO Care Management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Per member per month expenditures | 12 months

SECONDARY OUTCOMES:
Hospitalization days | 12 months
Outpatient visits | 12 months
Emergency Department visits | 12 months
Substance use disorder treatment | 12 months
Self-reported substance use | 12 months
Physical and mental functioning | 12 months
Depression | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: J Hunter Young, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- East Baltimore Medical Center, Baltimore, Maryland, United States